CLINICAL TRIAL: NCT02691832
Title: Measuring Core Body Temperature Using a Novel Non-invasive Sensor - a Follow up Study
Brief Title: Measuring Core Body Temperature Using a Novel Non-invasive Sensor
Acronym: Dräger
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-16-2920-HS-CTIL
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Body Temperature Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- research arm (Experimental): the trial contains one group which will undergo the described protocol three times:
  1. connected to rectal thermistor and to the double sensor
  2. connected to rectal thermistor, double sensor and cooling system of Icetron Technologies Ltd.
  3. connected to rectal thermistor and to the double sensor integrated into a helmet.
  Interventions: Device: "Dräger" double sensor

INTERVENTIONS:
Device: "Dräger" double sensor — The "Dräger" Double Sensor is a novel non-invasive device for assessing core body temperature.

SUMMARY:
The Double Sensor examined in this trial was developed by Dräger Company and is a novel non- invasive device for assessing core body temperature. In a preliminary research investigators have conducted the Double Sensor was found promising for potential use of physiological heat stress early detection. This follow-up experiment was designed to validate the data during high and changing body core temperatures and to examine the Double Sensor performance while integrated into a helmet as in intended application.

DETAILED DESCRIPTION:
12 healthy civilian volunteers will arrive to our lab and will undergo 4 experiment days: Recruitment day + VO2max test, 3 random days performing experiment protocol, dressed in uniforms: sitting in thermoneutral condition for one hour, afterwards they will walk on a treadmill in 5.5 km/h and 4% incline in hot chamber (40% celsius and 40% relative humidity) for 1.5 hours. Once connected to rectal thermistor and to the Double Sensor attached to the skin surface by sticker, once same as the day before with addition of cooling system of Icetron Technologies Ltd. worn on the wrist, and once connected to rectal thermistor and to the Double Sensor integrated into a helmet.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years.
* Healthy civilian volunteers.
* Without known medical illness or medication use.

Exclusion Criteria:

* History of heat injury.
* The existence or suspicion of existing cardiac or respiratory disease.
* Diabetes.
* Obesity.
* Infectious disease 3 days prior to the experiment.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Double sensor temperature | 3 days for each participant
  the Double Sensor will be attached to the forehead by sticker or integrated into a helmet. Double sensor temperature will be monitored continuously.
rectal temperature | 3 days for each participant
  rectal thermistor is the "gold standard" for core body temperature and will be measured continuously.

SECONDARY OUTCOMES:
heart rate | 4 days for each participant
  heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).
skin temperature | 3 days for each participant
  The skin temperature will be monitored by skin thermistors located at 3 sites (chest, arm and leg).

CONTACTS AND LOCATIONS:
Overall Officials: Haggai Schermann, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel

IPD SHARING:
Plan to Share IPD: No